CLINICAL TRIAL: NCT06958692
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial of Dextromethorphan and Bupropion Sustained-Release Tablets in Adult Patients With Major Depressive Disorder
Brief Title: A Trial of Dextromethorphan and Bupropion Sustained-Release Tablets in Patients With Major Depressive Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYH9052-002
Record Dates: First submitted 2025-03-30; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Dextromethorphan

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dextromethorphan and Bupropion (Experimental)
  Interventions: Drug: Dextromethorphan and Bupropion Sustained-Release Tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dextromethorphan and Bupropion Sustained-Release Tablets — Oral dextromethorphan and bupropion sustained-release tablets, taken daily for 6 weeks.
  Arms: Dextromethorphan and Bupropion
Drug: Placebo — Oral placebo tablets, taken daily for 6 weeks.
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, phase 3 trial, aim to evaluate the efficacy and safety of dextromethorphan and bupropion sustained-release tablets in Chinese adult patients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, Age 18 - 65, inclusive
2. Currently meets DSM-5 diagnosis of MDD without psychotic features, Current major depressive episode of at least 4 weeks in duration at screening
3. Identified as MDD by Mini-international Neuropsychiatric interview (M.I.N.I.)
4. MADRS score ≥25 and CGI-S ≥4 at screening and baseline
5. The results of physical examination and laboratory tests during the screening period meet the test requirements
6. Body Mass Index between 18 and 40 kg/m2, inclusive
7. For male subjects, use of an adequate method of birth control by the subject and by female sexual partners

Exclusion Criteria:

* 1. The researchers determined that it was refractory depression [defined as in a current depressive episode or a previous depressive episode, After 2 or more antidepressants, a sufficient amount (in the maximum recommendation of the manual), a course of foot therapy (at least even Continued medication for 4-6 weeks) ineffective after treatment] 2. The MADRS score improved by ≥ 25% at baseline compared with the screening period.

  3. Hospitalization in a psychiatric hospital during a current depressive episode 4. There is a clinically significant risk of suicide or self-harm and harm to others 5. Screening patients tested positive for substance abuse 6. In the investigator's judgment, there are any clinically significant oncology, hematology, or internal diseases that are not suitable for entry into the study Secretory/metabolic, cardiovascular, respiratory, kidney, liver, gastrointestinal, infectious or nervous system fever Or suffer from an unstable or progressive chronic disease 7. hypertension 8. Hypothyroidism or hyperthyroidism, except for the following cases: receiving stable medication with no change in dose for at least 1 month before screening (serum TSH must be > 0.75×LLN（ Lower Limit of Normal ） and < 1.25×ULN（Upper Limit of Normal ）) 9 Bupropion, dextromethorphan, opioids (such as codeine), or any of the study drugs Allergic to other ingredients 10. Presence of a history of intolerance to bupropion or dextromethorphan 11. People living with HIV, or testing positive for HIV during screening 12. Screening period hepatitis virology test positive 13. Liver enzyme test results during the screening period (total bilirubin, aspartate aminotransferase and/or alanine aminotransferase) > 2.0 × ULN 14. According to the investigator's judgment, other conditions are not suitable for participating in this clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in MADRS Total Score From Baseline to Week 6 | 6 weeks
  The MADRS is a 10-item scale and items are scored between 0-6 points. For each item, a score of 0 indicates the absence of symptoms, and a score of 6 indicates symptoms of maximum severity. A maximum total score is 60 points.

SECONDARY OUTCOMES:
Treatment response rate (the proportion of participants whose total score on the Montgomery-Åsberg Depression Rating Scale (MADRS) has improved by ≥ 50% compared to the baseline at the 6th week after administration) | 2 weeks
  The minimum MARDS score is 0, and the maximum score is 60. The higher the total score, the more severe the patient's depressive symptoms are.
Clinical cure rate (the proportion of participants with a total score of the Montgomery-Åsberg Depression Rating Scale (MADRS) ≤ 10 at the 2nd week after administration) | 6 weeks
  The minimum MARDS score is 0, and the maximum score is 60. The higher the total score, the more severe the patient's depressive symptoms are.
Proportion of participants with a ≥ 30% improvement in total MADRS scores from baseline at week 6 after administration | 6 weeks
  The minimum MARDS score is 0, and the maximum score is 60. The higher the total score, the more severe the patient's depressive symptoms are.
PGI-I score at week 6 after administration | 6 weeks
  （PGI-I：Patient Global Impression - Improvement）The minimum PGI-I score is 0, and the maximum score is 7 The higher the score, the more severe the degree of deterioration, while the lower the score, the better the improvement.
CGI-I score (Week 1, Week 2, Week 3, Week 4, Week 6) | 1，2，3，4，6 weeks
  CGI-I：Clinical Global Impressions - Improvement. The minimum CGI-I score is 1, and the maximum score is 7. The higher the score, the more severe the degree of deterioration, while the lower the score, the better the improvement.
Changes in CGI-S score from baseline to week 6 | 6 weeks
  CGI-S（Clinical Global Impressions-Severity）: The minimum CGI-S score is 0, and the maximum score is 7. The lower the score, the closer the patient's condition is to the normal state, while the higher the score, the more severe the condition.
Change in QIDS-SR-16 score from baseline to Week 6 | 6 weeks
  QIDS-SR-16（Quick Inventory of Depressive Symptomatology - Self-Report, 16-Item）：The minimum QIDS-SR-16 score is 0, and the maximum score is 27. The lower the score, the milder the depressive symptoms are, while the higher the score, the more severe the depressive symptoms are.
Change in SDS score from baseline to Week 6 | 6 weeks
  SDS（Self-Rating Depression Scale）：The minimum SDS score is 0, and the maximum score is 30. In the assessment, the lower the standard score, the milder the depressive state, and vice versa.
Incidence of adve rse events | Within 7 weeks
  Unit: % (proportion of participants experiencing adverse events to the total number of enrolled participants)
Incidence of serious adverse events | Within 7 weeks
  Unit: % (proportion of participants experiencing serious adverse events to the total number of enrolled participants)
Proportion of participants with significant abnormalities in vital signs | Within 7 weeks
  Unit: % (proportion of participants with significant vital sign abnormalities to the total number of enrolled participants)
  * Vital signs include:
  * Body temperature (axillary): ℃ (Celsius)
  * Respiration: times/minute
  * Pulse: times/minute
  * Sitting blood pressure: mmHg
Proportion of participants with significant abnormalities in physical examination results | Within 7 weeks
  * Unit: % (proportion of participants with significant physical examination abnormalities to the total number of enrolled participants)
  * Examination content includes: general condition, head and face, skin system, lymph nodes, eyes, ear-nose-throat, oral cavity, thyroid, respiratory system, cardiovascular system, abdomen, musculoskeletal system, nervous system, etc.
Proportion of participants with abnormal electrocardiogram (ECG) parameters | Within 7 weeks
  (The number of participants with significantly abnormal heart rate, respiratory rate (RR), PR interval, QRS duration, QT interval, and QTcF (in this study, the QT interval was corrected using Fridericia's formula).)
  o Unit: % (proportion of participants with abnormal ECG parameters to the total number of enrolled participants)
Proportion of participants with significant abnormalities in laboratory test results | Within 7 weeks
  o Unit: % (proportion of participants with significant laboratory test abnormalities to the total number of enrolled participants)
Incidence of suicidal ideation and behavior assessed by C-SSRS（Columbia Suicide Severity Rating Scale），It can comprehensively assess the individual's suicide risk level. The higher the score, the higher the suicide risk. | Within 7 weeks
  * Unit: % (proportion of participants with suicidal ideation or behavior to the total number of enrolled participants)
  * C-SSRS is a questionnaire used to evaluate participants' suicidal ideation and behavior, systematically assessing participants' suicidal status from three dimensions: suicidal ideation, intensity of ideation, and suicidal behavior.
Withdrawal responses as assessed by the PWC-20 | 7 weeks
  （Physician Withdrawal Checklist - 20）scale(The minimum PWC-20 score is 0, and the maximum score is 60. The higher the score, the more severe the condition.)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anding Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China